CLINICAL TRIAL: NCT05452135
Title: Investigation of Cognitive-Motor Dual Task and Swallowing Interaction in Healthy Young Adults
Brief Title: Cognitive - Motor Dual Task and Swallowing
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Other Study IDs: GO 22/417
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: DUAL TASK; DEGLUTİTİON; COGNİTİVE FUNCTİON; ACTİVİTİES OF DAİLY LİVİNG
Keywords: DUAL TASK; SWALLOW; COGNİTİVE; MOTOR FUNCTİONS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healty Adults: aged between 20 - 30 years right dominant being a volunteer to participate in the study
  Interventions: Other: Observation of visual, audotory and motor reaction time

INTERVENTIONS:
Other: Observation of visual, audotory and motor reaction time — Visual, auditory and motor reaction time will be measured as a result of the measurements made during the dual task evaluation.
  Other Names: Dual Task Assessment

SUMMARY:
Swallow and dual-task are a current issue and there are few studies on this subject. These studies have shown that as a result of dual-task interaction, swallowing is affected by attention and cognitive capacity, and dual-task negatively affects swallowing performance. But, studies include simple cognitive tasks and are not suitable for daily living activities. There is no study that compares all visual, auditory and motor dual tasks during swallowing and considers the effects on liquid, thick and solid foods similar to daily living activities. The aim of this study is to determine the effect of visual, auditory and motor dual-task on swallowing and chewing function in healthy young adults. As a result of the study, the dual-task that has the most impact on swallowing and chewing function will be determined, and visual, auditory and motor performance changes will be revealed as well as swallowing and chewing functions. It is planned that the results obtained will guide the rehabilitation of swallowing disorder with further studies on dual-task exercises.

DETAILED DESCRIPTION:
For many years, swallowing was thought of as a simple, reflexive activity controlled by the brainstem. However, studies on the neural control of swallowing have shown that cortical and subcortical structures of the nervous system are included in the neural control of swallowing, and swallowing consists of the pre-swallow phase, the oral preparatory phase, aoral phase, pharyngeal phase, and esophageal phase. And swallow prosses tarting with the perception of food.

Physical and chemical properties of the food, environmental factors, and motor, sensory and cognitive factors belonging to a person are effective in the swallowing process. Swallowing is an integral part of our daily life and we perform it together with other functions in our daily life. For example, while watching TV, in meetings, we continue to swallow/eat or drink. Even if we are not aware of swallowing, performing swallow and other functions at the same time. This situation called as "dual-task". 2 tasks performed at the same time always result in a decrease in the performance of one.

Swallow and dual-task are a current issue and there are few studies on this subject.These studies have shown that as a result of dual-task interaction, swallowing is affected by attention and cognitive capacity, and dual-task negatively affects swallowing performance. But, studies include simple cognitive tasks and are not suitable for daily living activities. There is no study that compares all visual, auditory and motor dual tasks during swallowing and considers the effects on liquid, thick and solid foods similar to daily living activities. The aim of this study is to determine the effect of visual, auditory and motor dual-task on swallowing and chewing function in healthy young adults. As a result of the study, the dual-task that has the most impact on swallowing and chewing function will be determined, and visual, auditory and motor performance changes will be revealed as well as swallowing and chewing functions. It is planned that the results obtained will guide the rehabilitation of swallowing disorder with further studies on dual-task exercises.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 - 30, being right dominant, be a volunteer to participate study

Exclusion Criteria:

* having a neurological disease

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: aged between 20- 30 healthy young adults.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-07-20 (Estimated); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
Dual Task assessment | 1 day
  Visual, auditory and motor reaction time will be measured as a result of the measurements made during the dual task evaluation.
Swallow assessment | 2 days
  During the dual task task, the dysphagia limit will be determined in liquid and viscous liquids. The maximum amount of water that the person can drink once will be used as the dysphagia limit.
Chewing Assessment | 2 days
  Participants will be asked to eat a 3x4 cm biscuit. Biscuit eating time, number of chewing cycles and number of bites will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Selen Serel Arslan, assoc. prof., Study Director — Hacettepe University Faculty of Physical Therapy and Rehabilitation Ankara, TURKEY

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Labeit B, Claus I, Muhle P, Regner L, Suntrup-Krueger S, Dziewas R, Warnecke T. Effect of cognitive and motor dual-task on oropharyngeal swallowing in Parkinson's disease. Eur J Neurol. 2021 Mar;28(3):754-762. doi: 10.1111/ene.14603. Epub 2020 Dec 2. PMID 33084118
- [Background] Shune SE, Moon JB. Effects of age and non-oropharyngeal proprioceptive and exteroceptive sensation on the magnitude of anticipatory mouth opening during eating. J Oral Rehabil. 2016 Sep;43(9):662-9. doi: 10.1111/joor.12419. Epub 2016 Jul 5. PMID 27377757